CLINICAL TRIAL: NCT05862363
Title: Small Intestinal Microbiota of Low Body Mass Index (BMI) & Normal BMI Women of Reproductive Age and Microbiota-directed Balanced Energy Protein (MD-BEP) Supplementation in Maternal Environmental Enteric Dysfunction (EED)
Brief Title: The Maternal EED Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Washington University School of Medicine (Other); Bangladesh Specialized Hospital (Unknown); Sheikh Russel National Gastroliver Institute & Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR-22117
Record Dates: First submitted 2023-02-08; First posted 2023-05-17 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Environmental Enteric Dysfunction (EED); Malnutrition; Women of Reproductive Age; Gut Microbiota; Balanced Energy Protein (BEP)
Keywords: Balanced energy protein (BEP); Environmental enteric dysfunction (EED); Gut microbiota; Malnutrition; Women of reproductive age
MeSH Terms: conditions — Malnutrition | interventions — Endoscopy, Digestive System; Counseling

STUDY DESIGN:
Intervention Model Description: All the activities in both Aim 1A and 1B are divided into two parallel arms. In 1A, EGD will be performed for both women within reproductive age with low-BMI and with normal-BMI. The interventions are designed in two arms. The first arm will enroll women from ages 18-35years with low BMI. They will be subdivided into two groups, each of which will receive either RUSF-BEP or MD-BEP. There will be cohort of healthy women with normal BMI for comparison. The second arm will consist of pregnant women from ages 18-35 years with low BMI. They will also be subdivided into two groups, each of which will receive either RUSF-BEP or MD-BEP. There will be cohort of healthy pregnant women with normal BMI for comparison.
Who Masked: Participant
Masking Description: The participants will be randomly assigned either RUSF or MDCF-2 (as dietary supplements). The participants will be made unaware of the supplement they are receiving; however, the field staff and investigators will be made aware of the dietary supplement allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Normal BMI women (Active Comparator): A total of 30 women with functional dyspepsia will be recruited as a control arm of AIM 1A. The women will be recruited who will present with GI symptoms. A total of 100 women will undergo EGD, out of which 30 women will be enrolled based on their diagnosis of functional dyspepsia and willingness to participate in the study.
  Interventions: Procedure: Esophagogastroduodenoscopy (EGD); Behavioral: Counselling and follow-up
- Low- BMI women (Active Comparator): A total of 60 women from low-socioeconomic status (SES) and with low BMI will be included in the intervention arm of aim A1. They will be recruited based on their willingness to participate and through meeting the inclusion criteria. They will under EGD, including collection of duodenal aspirates and 6-8 biopsy samples. After EGD, 30 participants will receive MD-BEP and 30 will receive RUSF-BEP upon randomization.
  Interventions: Dietary Supplement: Microbiota-directed balanced energy protein (MD-BEP); Dietary Supplement: Ready-to-use supplementary food-balanced energy protein (RUSF-BEP); Procedure: Esophagogastroduodenoscopy (EGD); Behavioral: Counselling and follow-up
- Low-BMI pregnant women (Active Comparator): We will recruit 60 pregnant women with low-BMI before 14 weeks of gestation. 30 participants will receive MD-BEP and 30 will receive RUSF-BEP upon randomization. They will be followed to note changes in weight gain, BMI, changes in EED biomarkers, gut microbial community repair, and pregnancy related outcomes.
  Interventions: Dietary Supplement: Microbiota-directed balanced energy protein (MD-BEP); Dietary Supplement: Ready-to-use supplementary food-balanced energy protein (RUSF-BEP); Behavioral: Counselling and follow-up
- Normal BMI pregnant women (Active Comparator): We will recruit 30 pregnant women with normal-BMI before 14 weeks of gestation. They will be provided with standard antenatal care. They will be followed to note changes in weight gain, BMI, changes in EED biomarkers, gut microbial community repair, and pregnancy related outcomes.
  Interventions: Behavioral: Counselling and follow-up

INTERVENTIONS:
Dietary Supplement: Microbiota-directed balanced energy protein (MD-BEP) — Prototypes for nutritional interventions that are composed of locally available, affordable, culturally acceptable complementary foods commonly consumed in Bangladesh have recently been developed.
  Arms: Low- BMI women; Low-BMI pregnant women
Dietary Supplement: Ready-to-use supplementary food-balanced energy protein (RUSF-BEP) — RUSF-BEP is composed of rice, lentil, sugar, soybean oil, and skimmed milk powder mixed with vitamin-mineral premix. MD-BEP is composed of chickpea flour, peanut flour, soy flour, green banana pulp, sugar, soybean oil, and vitamin-mineral premix. The results from previous studies support the notion that repair of impaired gut microbial community development could represent a new therapeutic concept for restoring healthy growth. RUSF-BEP will be given to one arm of low-BMI women of reproductive age and low-BMI pregnant women.
  Arms: Low- BMI women; Low-BMI pregnant women
Procedure: Esophagogastroduodenoscopy (EGD) — Aim 1A consists of performing EGD to women with low-BMI and normal BMI women with function dyspepsia. In order to enroll 30 participants with normal duodenal mucosal histology, we are planning to perform EGD on 100 healthy women (BMI 20-24.9 kg/m2) of childbearing age who have been referred for evaluation of functional dyspepsia. Undernourished low-BMI (<18.5kg/m2; 18-35 years) women of childbearing age will be enrolled from Bauniabadh and adjacent slum area of Mirpur, Dhaka and EGD will be performed among 60 women. A total of 6-8 biopsy samples from SI and a dry duodenal aspirate will be collected for biopsy, histochemical and immunocytochemical analysis.
  Arms: Low- BMI women; Normal BMI women
Behavioral: Counselling and follow-up — Normal BMI pregnant women will be counseled and followed up as per standard guidelines and will be provided routine antenatal care.

SUMMARY:
Undernutrition among women of reproductive age is more common in South Asia than in any other region. In South Asia, the prevalence of maternal undernutrition varies between 10 and 40%. There is a scarcity of data on the contribution of small intestinal (SI) microbiota to pathogenesis of Environmental Enteric Dysfunction (EED) of malnutrition, as it is difficult to obtain gut biopsy specimens from malnourished individuals, especially children. The Bangladesh Environmental Enteric Dysfunction (BEED) study, involving participants who live in an urban slum (Mirpur) in Dhaka, provided an opportunity to examine the role of the duodenal microbiota in the pathogenesis of EED in children and also performed esophagogastroduodenoscopy (EGD) on thirty-eight 18-45-year-old malnourished (BMI<18.5 kg/m2) women residing in the same resource-poor setting of Mirpur, Dhaka who failed to respond to an egg/milk/micronutrients- based nutritional intervention comparable to that given to children. In this intervention component, beginning at the end of the first trimester, low-BMI (<18.5 kg/m2) pregnant women (aged 18-35 years) will be randomly assigned to receive either Microbiota-directed Balanced Energy Protein (MD-BEP) or Ready-to-Use-Supplementary Food Balanced Energy Protein (RUSF-BEP) for the duration of their pregnancy and during the first 3 postnatal months, in addition to standard antenatal care. A parallel cohort of age-matched normal-BMI pregnant women who will not receive any nutritional intervention will serve as a reference control group.

DETAILED DESCRIPTION:
Specific Objectives:

AIM 1 - Human studies component Comparative assessment of low BMI & normal BMI small intestinal (SI) and fecal microbiomes plus feature of SI mucosal, plasma and fecal proteomes prior to intervention.

Intervention with MD-BEP to access effect on EED microbiome and physiologic state of low BMI women.

Identify candidate mediators/surrogate biomarkers of EED (fecal/plasma) that can be deployed in future clinical studies.

AIM 1A will compare the SI and fecal microbiota and the plasma, duodenal and fecal proteomes/ metabolomes of non-pregnant, young malnourished Bangladeshi women (BMI<18.5kg/m2) who have histopathologic evidence of SI enteropathy versus those with normal BMIs (20-24.9kg/m2) and no histopathologic evidence of enteropathy who have undergone routine endoscopic evaluation for dyspepsia.

AIM 1B The investigators will perform an intervention study, beginning at the end of the first trimester, in which low-BMI (<18.5 kg/m2) pregnant women (aged 18-35 years) will be randomly assigned to receive either MD-BEP or RUSF-BEP for the duration of their pregnancy and during the first 3 postnatal months, in addition to standard antenatal care (n=30/arm). A parallel cohort of age-matched normal-BMI pregnant women who will not receive any nutritional intervention will serve as a reference control group.

AIM 2 - Preclinical Component This Aim has two parts - a therapeutic target identification component (AIM 2A) and a glycan therapeutic development component (AIM 2B).

Test of MD-BEP and new maternal microbiome directed glycans to ameliorate enteropathy/Biomarker of EED.

Background of the Project including Preliminary Observations:

Undernutrition among women of reproductive age is more common in South Asia than in any other region. In South Asia, the prevalence of maternal undernutrition varies between 10 and 40%. Particularly in Bangladesh, the prevalence of undernutrition among women is much higher than in any other developing country, with more than 30% of women of reproductive age reported to be malnourished. Maternal undernutrition has persistently been described to be a major contributor to child morbidity, mortality, and poor birth outcomes, including low birth weight (LBW), neonatal mortality, and subsequent childhood undernutrition. Maternal undernutrition alone accounts for about 25-50% of intrauterine growth restriction. In such a way, under-nutrition can be transferred from one generation to other. Half of the under-five children in slums of Bangladesh are stunted having retarded linear growth compared to one-third in non-slum areas.

The prevention or treatment of intergenerational malnutrition represents a critical medical need that is yet to be addressed and remains a pressing global health challenge. There is a scarcity of data on the contribution of small intestinal (SI) microbiota to pathogenesis of Environmental Enteric Dysfunction (EED) of malnutrition, as it is difficult to obtain gut biopsy specimens from malnourished individuals, especially children. The Bangladesh Environmental Enteric Dysfunction (BEED) study, involving participants who live in an urban slum (Mirpur) in Dhaka, provided an opportunity to examine the role of the duodenal microbiota in the pathogenesis of EED in children and also performed esophagogastroduodenoscopy (EGD) on thirty-eight 18-45-year-old malnourished (BMI<18.5 kg/m2) women residing in the same resource-poor setting of Mirpur, Dhaka who failed to respond to a egg/milk/micronutrients- based nutritional intervention comparable to that given to children. It was observed that malnourished women of childbearing age living in Mirpur exhibit small intestinal enteropathy resembling that found in Mirpur children with EED. In this proposal, our primary aim is to test the hypothesis that the SI microbiota contributes to SI enteropathy and malnutrition (low-BMI) in young Bangladeshi women of childbearing age. Furthermore, there is some initial evidence that pregnancy outcomes can be predicted by the features of the gut microbiota of pregnant women. The maternal gut microbiota itself may influence the development of the offspring cohort, both in prenatal and postnatal life. As maternal gut microbiota, directly and indirectly, influences the metabolism of the fetus and infants, it may be possible to optimize gestational weight gain (GWG), pregnancy outcomes, and subsequent growth and development of children through modulation of intestinal microbiota in women during pregnancy and lactation. Therefore, a corollary of our primary aim is that direct or indirect transmission of the gut microbiota of mothers with EED to their children perpetuates intergenerational undernutrition.

Conventional nutritional interventions or low-cost water and sanitation interventions may be ineffective in reversing EED-related growth faltering in children, warranting microbiota/microbiome targeted food and other interventions. Prototypes for nutritional interventions that are composed of locally available, affordable, culturally acceptable complementary foods commonly consumed in Bangladesh have recently been developed. Microbiota- directed complementary food (MDCF) formulations were subsequently tested in a pre-proof-of-concept (POC) study involving 12-18-month-old Bangladeshi children with moderate acute malnutrition (MAM) living in the same slum (Mirpur). One of the MDCFs, MDCF-2, was distinguished from the other formulations based on its superior performance based on certain parameters including growth.

The latest WHO antenatal care guideline advises implementing balanced energy and protein (BEP) supplementation for pregnant women residing in undernourished communities. The Bill and Melinda Gates Foundation organized an expert consultation in September 2016 to develop nutrient content targets for affordable nutritional supplements for pregnant and lactating women in undernourished settings. The expert consultation recommended that women in undernourished settings receive a daily BEP supplement containing 250-500 kcal of energy and 14-18 grams of protein. With this in mind, we propose to include an interventional component involving the administration of microbiota-directed balanced energy protein (MD-BEP) in pregnant and non-pregnant low-BMI women. This modified BEP will contain ingredients from the previously mentioned MDCF-2 that are aimed at improving microbiota. With this in mind, the investigators propose to include an interventional component involving the administration of MD-BEP in pregnant and non-pregnant low-BMI women. In this intervention component, beginning at the end of the first trimester, low-BMI (<18.5 kg/m2) pregnant women (aged 18-35 years) will be randomly assigned to receive either the MD-BEP or Ready-use-supplementary food-balanced energy protein (RUSF-BEP) for the duration of their pregnancy and during the first three postnatal months, in addition to standard antenatal care. A parallel cohort of age-matched normal-BMI pregnant women who will not receive any nutritional intervention will serve as a reference control group. In this intervention component, beginning at the end of the first trimester, low-BMI (<18.5 kg/m2) pregnant women (aged 18-35 years) will be randomly assigned to receive either the MD-BEP or RUSF-BEP for the duration of their pregnancy and during the first 3 postnatal months, in addition to standard antenatal care. A parallel cohort of age-matched normal-BMI pregnant women who will not receive any nutritional intervention will serve as a reference control group.

The investigators will test the hypothesis that small intestinal microbiota contributes to small intestinal enteropathy and malnutrition in young Bangladeshi women of childbearing age. An interventional component will be included involving the administration of MD-BEP in pregnant and non-pregnant low-BMI women. This will be based on the hypothesis that transmission of the microbiota of mothers with EED to their children perpetuates intergenerational undernutrition.

The overarching goals for the current study will be to:

1. Delineate mechanisms by which the SI microbial community obtained from low-BMI Mirpur women contributes to maternal malnutrition and identify surrogate biomarkers that can be applied to malnourished pregnant women
2. Test whether MD-BEP can ameliorate EED as judged by these surrogate endpoints in low-BMI women (who are either pregnant or non-pregnant)
3. Develop a gnotobiotic mouse model of maternal EED using culture collections from malnourished low-BMI as well as normal BMI women, and identify microbial therapeutic targets in their SI microbiota, and
4. Perform preclinical tests of MD-BEP and candidate therapeutic glycans in gnotobiotic mice to identify/develop candidate glycan/synbiotic therapeutics for future clinical studies. These preclinical models will also serve as a platform for testing candidate therapeutics arising from other BMGF-sponsored initiatives where there is good confidence in rationale.

To achieve the goals, in this proposed study the investigators will use two specific aims involving the human subjects, AIM 1A and AIM 1B. In AIM 1A the investigators will compare the SI and fecal microbiota and the plasma, duodenal and fecal proteomes/ metabolomes of non-pregnant, young malnourished Bangladeshi women (BMI<18.5kg/m2) who have histopathologic evidence of SI enteropathy versus those with normal BMIs (20-24.9kg/m2) and no histopathologic evidence of enteropathy who have undergone routine endoscopic evaluation for dyspepsia. In AIM 1B, the investigators will perform an intervention study, beginning at the end of the first trimester, in which low-BMI (<18.5 kg/m2) pregnant women (aged 18-35 years) will be randomly assigned to receive either MD-BEP or RUSF-BEP for the duration of their pregnancy and during the first 3 postnatal months, in addition to standard antenatal care (n=30/ arm). A parallel cohort of age-matched normal-BMI pregnant women who will not receive any nutritional intervention will serve as a reference control group.

Methods:

In AIM 1A, for the healthy group, the investigators plan to recruit a cohort of normal-BMI Bangladeshi women who will undergo esophagogastroduodenoscopy (EGD) for evaluation of functional dyspepsia and our goal is to identify 30 normal BMI participants who have normal duodenal mucosal histology and collect duodenal biopsies, duodenal aspirates, plus plasma and fecal specimens from these participants at the time of endoscopy. In order to enroll these 30 participants with normal duodenal mucosal histology, the investigators are planning to perform EGD on 100 healthy women (BMI 20-24.9 kg/m2) of childbearing age who have been referred for evaluation of functional dyspepsia. Participants will be screened from women attending Gastroenterology OPD of Sheikh Russel National Gastroliver Institute and Hospital, the Bangladesh Specialized Hospital, Dhaka, Bangladesh, and the community, who meet the inclusion criteria.

Undernourished low-BMI (<18.5kg/m2; 18-35 years) women of childbearing age will be enrolled from Bauniabadh and adjacent slum area of Mirpur, Dhaka and EGD will be performed among 60 women at icddr,b Dhaka Hospital, Sheikh Russel National Gastroliver Institute and Hospital, Bangladesh Specialized Hospital, or icddr,b hospital, Dhaka. Participants will be screened through household surveys from the Bauniabadh and adjacent slum area of from Mirpur, Dhaka. The endoscopist is the same individual who performed EGD on the children as well as malnourished women in the BEED study. After EGD, the low-BMI women will be randomized into two groups and receive daily dietary supplementation with either MD-BEP or RUSF-BEP for a period of 90 days, with a further 270 days of follow-up after cessation of the intervention and biological samples will be collected from the participants according to the schedule. Healthy women with normal BMI who underwent EGD will also be followed similarly for 360 days, without any nutritional intervention.

A nested sub-study will be done under aim 1A to test the Small Intestine MicroBiome Aspiration (SIMBA) capsule, a small, ingestible pill that can selectively sample the small intestine microbiome. The SIMBA study will apply for approval through a separate protocol. For AIM 1B, beginning at the end of the first trimester, in which low-BMI (<18.5 kg/m2) pregnant women (aged 18-35 years) will be randomly assigned to receive either MD-BEP or RUSF-BEP for the duration of their pregnancy and during the first 3 postnatal months, in addition to standard antenatal care (n=30/arm). A parallel cohort of age-matched normal-BMI pregnant women who will not receive any nutritional intervention will serve as a reference control group. The investigators are planning to test a minimal-risk device to collect tissue samples from the small intestine (e.g. trans- nasal introduction tube or TNIT) in a sub-sample of pregnant women under our Aim 1b of our proposed proposal. Therefore, a nested sub-study will be done under aim 1B to test tethered capsule endoscopy (TNIT) to study small- intestinal morphology for EED in a group of 15 pregnant women enrolled in the study based on the assumption that by the time this technology would be validated with conventional endoscopy in women of reproductive age under the Experimental Medicine Platform (Protocol # PR-22082) as well as safety data will be available on pregnant women from the study conducted elsewhere. The participants of this sub-study will be selected randomly from those who will provide their consent to participate in the sub-study. In addition, a preclinical component will be performed aimed at a therapeutic target identification component (AIM 2A) and a glycan therapeutic development objective (AIM 2B) at Washington University in St. Louis.

The investigators plan to recruit a cohort of normal-BMI Bangladeshi women who will undergo esophagogastroduodenoscopy (EGD) for evaluation of functional dyspepsia and our goal is to identify 30 normal BMI participants who have normal duodenal mucosal histology and collect duodenal biopsies, duodenal aspirates, plus plasma and fecal specimens from these participants at the time of endoscopy. Moreover, plasma and fecal samples will be collected according to the follow-up schedule.

Sites:

Participants will be screened from those attending gastroenterology out-patient department (OPD) of Sheikh Russel National Gastroliver Institute and Hospital Bangladesh Specialized Hospital, and from the community who meet the inclusion criteria.

Field Site:

Participants will be screened through household surveys from the Bauniabadh and adjacent slum area of from Mirpur, Dhaka (Fig.4). This area is densely populated and is located 7-8 km from the icddr,b Dhaka Hospital at Mohakhali. Mirpur is selected as the study site because it is inhabited by poor and middle- class families, residential and sanitary conditions are typical of any congested urban settlement, and the study investigators have ongoing research activities in the area. The site has a typical squatter settlement; the average family size of households is 4.5, with 48% females. About 20% of households have a monthly income of only US$62, 30% of mothers never attended school, and only 3% obtained secondary school education. The majority of the people are day laborers, garment workers, and transport workers. Mirpur has a population of about half a million in an area of 14.22 km2. More than 38, 000 people live in each square kilometer of the area compared with the mean of 8229/km2 in Dhaka district and 976/km2 in Bangladesh17.

Screening, recruitment and consenting Census, screening, enrolment of subjects (low-BMI women) will be done in Bauniabadh area of Mirpur in Dhaka city. Women who meet the inclusion-exclusion criteria will be approached about enrolment into this study. A trained Field Research Assistant (FRA) will explain the study in detail, answer any questions from the participant or her relatives, and invite her for enrolment in the study. If she is interested to volunteer in the study, the designated staff will proceed to screening and consenting.

Screening will consist of a review of the inclusion and exclusion criteria listed above. A detailed history will be obtained from the participants following clinical examination. Adult participants who fulfill the inclusion criteria and are not excluded through history and clinical examination will undergo following screening tests based on clinical judgement: Chest x-ray, urine for R/E, ultrasonography of whole abdomen, fasting blood glucose/ HbA1c, stool for occult blood test (OBT), cancer markers (ie. CEA, CA 15.3, CA 19.9). Patients diagnosed with any abnormal lab test results will be treated by the study physician as per standard guidelines. Patients requiring expert opinion regarding any complicated clinical condition will be referred to a subject specialist accordingly.

If the subject is eligible to participate, the process will proceed to consenting, consisting of a thorough review of the written consent form in a manner appropriate for their literacy level. Prior to signing the consent form, she will have an opportunity to ask any questions about the study. If the FRA determines that participants have demonstrated adequate comprehension of the study, the consent form will be signed by the FRA and the participant. If the participant is not sufficiently literate to read and/or sign the consent form, consenting and a thumbprint signature will be obtained in the presence of a witness who is not associated with the study. The participant will be provided with a copy of the signed consent form.

EGD and biopsy sample collection Endoscopy will be performed at the Sheikh Rasel Gastro Liver Institute and Hospital and the Bangladesh Specialized Hospital. The endoscopist is the same individual who performed EGD on the children as well as malnourished women in the BEED study. Clinical metadata will be collected, including socio-demographic data, dietary history, and use of antibiotics and proton pump inhibitors (PPI) during 12-months prior to EGD [note that consumption of PPIs is common in Bangladesh; in one representative study of an outpatient clinic population the incidence was 72%, with >30% of individuals obtaining PPIs without a prescription]. A tissue transglutaminase (tTG) test will be used to rule out Celiac Disease.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for pregnant low-BMI women

1. Bangladeshi female, age 18-35 years
2. BMI 20-24.9 kg/m2
3. Middle-upper socioeconomic class (≥ $11/day family income)
4. Functional dyspepsia
5. Willing to sign the consent form
6. Willing to provide biological samples during the study period of 6 months

Inclusion criteria for non-pregnant low-BMI women 1. Bangladeshi female, age 18-35 years

1. BMI <18.5 kg/m2
2. No antibiotics for 1 month
3. Willing to sign the consent form
4. Willing to undergo endoscopy and biopsy
5. Willing to provide biological samples during the study period of 6 months
6. Willing to receive food supplementation for 3 months

Inclusion criteria for normal-BMI non-pregnant women

1. Bangladeshi female, age 18-35 years
2. BMI 20-24.9 kg/m2
3. Middle-upper socioeconomic class (≥ $11/day family income)
4. Functional dyspepsia
5. Willing to sign the consent form
6. Willing to provide biological samples during the study period of 6 months

Inclusion criteria for normal-BMI pregnant women

1. Bangladeshi female, age 18-35 years
2. BMI 20-24.9 kg/m2
3. Middle-upper socio-economic class (≥ $11/day family income)
4. Enrolled at the end of first-trimester of pregnancy (before 14 weeks of gestation)
5. Willing to sign the consent form
6. Willing to undergo endoscopy and biopsy
7. Willing to provide biological samples during the study period
8. Willing to let anthropometry and biological sample collection from her newborn for the first 6 months of life

Exclusion Criteria:

Exclusion criteria for pregnant low-BMI women

1. Received antibiotics during the last one month
2. Presence of any chronic disease including diabetes mellitus or any congenital disorder or deformity
3. Ongoing episode of diarrhea, history of persistent diarrhea in the past month or history of acute diarrhea in the past 7 days

Exclusion criteria for non-pregnant low-BMI women

1. Severe anemia (<8 g/dl), TB and other chronic diseases, including diabetes mellitus, urogenital infections or any congenital disorder or deformity
2. Pregnancy, lactation, drug abuse, known psychiatric disorders
3. High clinical suspicion of cancer or other chronic or acute diseases that may cause malnutrition. Adult participants who fulfill the inclusion criteria and are not excluded through history and clinical examination will undergo following screening tests based on clinical judgement:

   1. Chest x-ray
   2. Urine for R/E
   3. Ultrasonography of whole abdomen
   4. Fasting blood glucose/ HbA1c
   5. Stool for OBT (occult blood test)
   6. Cancer markers (ie. CEA, CA 15.3, CA 19.9)
4. Known allergy to any components of nutrition intervention
5. Nugent Score/Amsel Criteria to exclude bacterial vaginosis: A Nugent score 3-4 is consistent with Bacterial vaginosis (BV). The modified Amsel criteria with a cut-off value of 2 (pH+VD; sensitivity 71%, specificity 90%, accuracy 88% or KOH+VD; sensitivity 75%, specificity 91%, accuracy 89%) might be considered for this purpose20.
6. Ongoing episode of diarrhea, history of persistent diarrhea in the past month or history of acute diarrhea in the past 7 days

Exclusion criteria for non-pregnant normal-BMI women

1. Received antibiotics during the last one month
2. Presence of any chronic disease including diabetes mellitus or any congenital disorder or deformity
3. Ongoing episode of diarrhea, history of persistent diarrhea in the past month or history of acute diarrhea in the past 7 days

Exclusion criteria for pregnant normal-BMI women

1. Multiple pregnancy (carrying two or more fetuses)
2. Threatened abortion, persistent pervaginal bleeding, or cervical incompetence
3. History of three or more consecutive abortions
4. History of gestational diabetes, macrosomia, gestational hypertension, preeclampsia/eclampsia in a prior pregnancy
5. Active disease/complications requiring acute phase treatment in a hospital
6. Tuberculosis
7. Severe anemia (Hb concentration < 8 mg/dl)
8. Antibiotic use (ongoing or within last two weeks before the onset of intervention)
9. Taking medications such as insulin, thyroid hormones, glucocorticoids
10. Chronic diseases, such as hypertension, heart disease, chronic obstructive pulmonary disease, chronic kidney disease, chronic liver disease, pancreatic diseases, Crohn's disease, ulcerative colitis, diabetes mellitus, thyroid dysfunction, immunological diseases, malignancy, or any congenital disorder or other diseases which could impede compliance with the study protocol
11. Known case of serious psychiatric or behavioral disorders, such as schizophrenia, bipolar disorder
12. Having known history of allergy to the therapeutic agents
13. Having a plan to move or deliver outside the study area
14. Known allergy to any components of nutrition intervention.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — For this study, we will enroll pregnant women and non-pregnant women of reproductive age with low-BMI. They will be compared with a matched cohort of women with normal BMI. The women will be within reproductive age.
Enrollment: 180 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of weight in women of reproductive age before and after nutritional intervention | Enrolment to 360 days for non-pregnant cohort, and up to 540 days for pregnant cohort
  In this study, nutritional status will be assessed through anthropometry. Body weight will be collected in kg using a standard weighing machine, and determined at the time of enrolment for all groups, days 30, 60, 90, 120, 180, 210, 270, and 360 for non-pregnant cohort; and days 30, 60, 90, 120, 164, 178, 180, 210, 280, 360, 390, 450, and 540 for pregnant cohort.
Height of women of reproductive age before and after nutritional intervention | Enrolment to 360 days for non-pregnant cohort, and up to 540 days for pregnant cohort
  In this study, nutritional status will be assessed through anthropometry. Height will be collected in centimeters using stadiometer. Anthropometry will be collected at the time of enrolment for all groups, days 30, 60, 90, 120, 180, 210, 270, and 360 for non-pregnant cohort; and days 30, 60, 90, 120, 164, 178, 180, 210, 280, 360, 390, 450, and 540 for pregnant cohort.
Change in BMI of women of reproductive age before and after nutritional intervention | Enrolment to 360 days for non-pregnant cohort, and up to 540 days for pregnant cohort
  In this study, nutritional status will be assessed through anthropometry. Body weight in kilogram and height in cm will be determined at the time of enrolment for all groups, days 30, 60, 90, 120, 180, 210, 270, and 360 for non-pregnant cohort; and days 30, 60, 90, 120, 164, 178, 180, 210, 280, 360, 390, 450, and 540 for pregnant cohort.
Change in body composition of total fat and fat-free mass of women of reproductive age before and after nutritional intervention before and after nutritional intervention | Enrolment to 360 days for non-pregnant, up to 540 days for pregnant cohort
  Bioelectric Impedance Analysis (BIA) will be used to measure total fat and fat-free mass before, during and after the intervention. BIA is a method of assessing the body composition by measuring the body fat in relation to lean body mass. It is an integral part of a health and nutrition assessment. BIA will be used to measure total fat and fat-free mass before and after intervention with each of the three arms. 60 low-BMI women (18-35 years) provided with MD-BEP/RUSF-BEP intervention, with an age-matched cohort of 30 healthy (normal-BMI) women and subsequent serial fecal and plasma sampling (without nutritional intervention) serving as a control group will be selected for this analysis. Data will be collected on days 1, 180, and 360 days for non-pregnant women and days 0, 180, 360, and 540 days for pregnant women, and the unit of measurement will be the percentage of fat.
Validated plasma biomarker (sCD14) | Enrolment to 360 days for non-pregnant and children, up to 540 days for pregnant cohort
  Blood will be collected at enrolment, and days 30, 90, 180, 270, 360 for non-pregnant women; days 0, 30, 90, 180, 270, 360, 450, and 540 for pregnant women; and days 30, 180, 270, and 360 for offspring cohort, , to determine changes in the representation of plasma biomarkers of EED as a function of treatment. Plasma sCD14 will be measured by ELISA method and it serves as a marker for Systemic inflammation
Validated plasma biomarker (CRP) | Enrolment to 360 days for non-pregnant and children, up to 540 days for pregnant cohort
  Blood will be collected at enrolment and on days 30, 90, 180, 270, 360 for non-pregnant women; days 0, 30, 90, 180, 270, 360, 450, and 540 for pregnant women; and days 30, 180, 270, and 360 for the offspring cohort to determine changes in the representation of plasma biomarkers of EED as a function of treatment. Plasma c-reactive protein (CRP) will be measured by the ELISA method.
Validated plasma biomarker (AGP) | Enrolment to 360 days for non-pregnant and children, up to 540 days for pregnant cohort
  Blood will be collected at enrolment, and days 30, 90, 180, 270, 360 for non-pregnant women; days 0, 30, 90, 180, 270, 360, 450, and 540 for pregnant women; and days 30, 180, 270, and 360 for offspring cohort, to determine changes in the representation of plasma biomarkers of EED as a function of treatment. alpha-1-acid glycoprotein (AGP) will serve as a marker for Systemic inflammation and it will be measured by ELISA method.
Hormonal regulators of appetite and satiety (Leptin) | Enrolment to 360 days for non-pregnant and children, up to 540 days for pregnant cohort
  Blood will be collected at enrolment, and days 30, 90, 180, 270, 360 for non-pregnant women; days 0, 30, 90, 180, 270, 360, 450, and 540 for pregnant women; and days 30, 180, 270, and 360 for offspring cohort, to determine changes in the representation of plasma biomarkers of EED as a function of treatment. Leptin will serve as a marker for Hormonal regulators of appetite and satiety and it will be measured by ELISA method from plasma.
Hormonal regulators of appetite and satiety (Ghrelin) | Enrolment to 360 days for non-pregnant and children, up to 540 days for pregnant cohort
  Blood will be collected at enrolment, and days 30, 90, 180, 270, 360 for non-pregnant women; days 0, 30, 90, 180, 270, 360, 450, and 540 for pregnant women; and days 30, 180, 270, and 360 for offspring cohort, , to determine changes in the representation of plasma biomarkers of EED as a function of treatment. Ghrelin will serve as a marker for Hormonal regulators of appetite and it will be measured by ELISA method from Plasma.
Hormonal regulators of appetite and satiety (IGF-1) | Enrolment to 360 days for non-pregnant and children, up to 540 days for pregnant cohort
  Blood will be collected at enrolment, and days 30, 90, 180, 270, 360 for non-pregnant women; days 0, 30, 90, 180, 270, 360, 450, and 540 for pregnant women; and days 30, 180, 270, and 360 for offspring cohort, , to determine changes in the representation of plasma biomarkers of EED as a function of treatment. Insulin-like growth factor 1 (IGF-1) will serve as a marker for Hormonal regulators of appetite and satiety and it will be measured from plasma using ELISA method.
Hormonal regulators of appetite and satiety (Glucagon-like peptide-2 (GLP-2)) | Enrolment to 360 days for non-pregnant and children, up to 540 days for pregnant cohort
  Blood will be collected at enrolment, and days 30, 90, 180, 270, 360 for non-pregnant women; days 0, 30, 90, 180, 270, 360, 450, and 540 for pregnant women; and days 30, 180, 270, and 360 for offspring cohort,, to determine changes in the representation of plasma biomarkers of EED as a function of treatment. Glucagon-like peptide-2 (GLP-2)will serve as a marker for Hormonal regulators of appetite and satiety and it will be measured from plasma using ELISA method.
Micronutrients level in plasma (Ferritin) | Enrolment to 360 days for non-pregnant and children, up to 540 days for pregnant cohort
  Blood will be collected at baseline (at the time of EGD),enrolment, and days 30, 90 and, 180, 270, 360 for non-pregnant women; days 0, 30, 90, 180, 270, 360, 450, and 540 for pregnant women; and days 30, 180, 270, and 360 for offspring cohort,, to determine changes in the representation of plasma biomarkers of EED as a function of treatment. Ferritin will serve as a marker for micronutrient level in the blood and it will be measured by ELISA method from Plasma.
Micronutrients level in plasma (Zinc) | Enrolment to 360 days for non-pregnant and children, up to 540 days for pregnant cohort
  Blood will be collected at baseline (at the time of EGD),enrolment, and days 30, 90 and, 180, 270, 360 for non-pregnant women; days 0, 30, 90, 180, 270, 360, 450, and 540 for pregnant women; and days 30, 180, 270, and 360 for offspring cohort,, to determine changes in the representation of plasma biomarkers of EED as a function of treatment. Zinc will serve as a marker for micronutrient level in the blood and the plasma zinc will be measured by atomic absorption spectrometry method.
Validated fecal biomarkers of health status including mediators of growth, systemic inflammation, gut inflammation/enteropathogenic burden, stool pH | Enrolment to 360 days for non-pregnant and children, up to 540 days for pregnant cohort
  Fecal samples will be collected at the time Of enrolment, days 30, 60, 90, 120, 180, 210, 270, 360 for non-pregnant women; days 0, 30, 60, 90, 120, 180, 210, 270, 360, 390, 450, and 540 for pregnant women; and days 0, 30, 90, 180, 210, 270, and 360 for offspring cohort, of enrolment, days 30, 60, 90, 120, 180, 210, 270, 360 for non-pregnant women; days 0, 30, 60, 90, 120, 180, 210, 270, 360, 390, 450, and 540 for pregnant women; and days 0, 30, 90, 180, 210, 270, and 360 for offspring cohort, for analysis of the effects of intervention on the microbiota-microbiome. Stool pH will be measured on freshly collected stool samples by portable stool pH meter from Hanna instruments, USA.
15. Validated fecal biomarkers of health status including mediators of growth, systemic inflammation, gut inflammation/ enteropathogenic burden) (Myeloperoxidase) | Enrolment to 360 days for non-pregnant and children, up to 540 days for pregnant cohort
  Fecal samples will be collected at the time of enrolment, days 30, 60, 90, 120, 180, 210, 270, 360 for non-pregnant women; days 0, 30, 60, 90, 120, 180, 210, 270, 360, 390, 450, and 540 for pregnant women; and days 0, 30, 90, 180, 210, 270, and 360 for offspring cohort, for analysis of the effects of intervention on the microbiota-microbiome. Myeloperoxidase will be measured from fecal samples using ELISA method.
Validated fecal biomarkers of health status including mediators of growth, systemic inflammation, gut inflammation/enteropathogenic burden (neopterin) | Enrolment to 360 days for non-pregnant and children, up to 540 days for pregnant cohort
  Fecal samples will be collected at the time of enrolment, days 30, 60, 90, 120, 180, 210, 270, 360 for non-pregnant women; days 0, 30, 60, 90, 120, 180, 210, 270, 360, 390, 450, and 540 for pregnant women; and days 0, 30, 90, 180, 210, 270, and 360 for offspring cohort, for analysis of the effects of intervention on the microbiota-microbiome. Neopterin will be measured from fecal sample using ELISA method
Validated fecal biomarkers of health status including mediators of growth, systemic inflammation, gut inflammation/enteropathogenic burden (calprotectin) | Enrolment to 360 days for non-pregnant and children, up to 540 days for pregnant cohort
  Fecal samples will be collected at the time of enrolment, days 30, 60, 90, 120, 180, 210, 270, 360 for non-pregnant women; days 0, 30, 60, 90, 120, 180, 210, 270, 360, 390, 450, and 540 for pregnant women; and days 0, 30, 90, 180, 210, 270, and 360 for offspring cohort, for analysis of the effects of intervention on the microbiota-microbiome. Calprotectin will be measured from fecal sample using ELISA method.
Validated fecal biomarkers of health status including mediators of growth, systemic inflammation, gut inflammation/enteropathogenic burden (Dual oxidase 2 (DUOX2) | Enrolment to 360 days for non-pregnant and children, up to 540 days for pregnant cohort
  Fecal samples will be collected at the time of enrolment, days 30, 60, 90, 120, 180, 210, 270, 360 for non-pregnant women; days 0, 30, 60, 90, 120, 180, 210, 270, 360, 390, 450, and 540 for pregnant women; and days 0, 30, 90, 180, 210, 270, and 360 for offspring cohort, for analysis of the effects of intervention on the microbiota-microbiome. Fecal DUOX2 will be measured by ELISA method.
Validated fecal biomarkers of health status including mediators of growth, systemic inflammation, gut inflammation/enteropathogenic burden (Oxidation-Reduction Potential (Redox potential)) | Enrolment to 360 days for non-pregnant and children, up to 540 days for pregnant cohort
  Fecal samples will be collected at the time of enrolment, days 30, 60, 90, 120, 180, 210, 270, 360 for non-pregnant women; days 0, 30, 60, 90, 120, 180, 210, 270, 360, 390, 450, and 540 for pregnant women; and days 0, 30, 90, 180, 210, 270, and 360 for offspring cohort, for analysis of the effects of intervention on the microbiota-microbiome. Redox potential will be measured in millivolt (mV)
Validated fecal biomarkers of health status including mediators of growth, systemic inflammation, gut inflammation/enteropathogenic burden Lipocalin 2 (Lcn2) | Enrolment to 360 days for non-pregnant and children, up to 540 days for pregnant cohort
  Fecal samples will be collected at the time of enrolment, days 30, 60, 90, 120, 180, 210, 270, 360 for non-pregnant women; days 0, 30, 60, 90, 120, 180, 210, 270, 360, 390, 450, and 540 for pregnant women; and days 0, 30, 90, 180, 210, 270, and 360 for offspring cohort, for analysis of the effects of intervention on the microbiota-microbiome. Lipocalin 2 (Lcn2) will be measured by ELISA method using fecal sample.
Pregnancy-related change in weight | Enrolment to pregnancy termination and three months post-birth
  Pregnant women will be enrolled and followed up over a period of 9 months. Enrolment will be done before 2nd trimester. Low-BMI pregnant women will be provided with daily supplementation of supplemental food (MD-BEP/RUSF-BEP) and normal-BMI women will be followed without any intervention. For the low-BMI pregnant women, antenatal care (ANC) services from nearby healthcare facility will be ensured by study staff. Trained Health Workers (HWs) will visit the homes of all enrolled pregnant women once a month. During the follow up, the investigators will collect anthropometry data from each participant every four-weekly. The unit of data collection for pregnant women is kg. Relevant laboratory investigation that will be done among pregnant women will follow previously described methods.

CONTACTS AND LOCATIONS:
Overall Officials: Md. Shabab Hossain, MBBS, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b), Dhaka, Dhaka Division, Bangladesh

IPD SHARING:
Plan to Share IPD: No